CLINICAL TRIAL: NCT00940758
Title: Phase I and Pharmacokinetic Study of Biweekly PEP02 (Liposome Irinotecan) in Patients With Metastatic Colorectal Cancer Refractory to First-line Oxaliplatin-based Chemotherapy
Brief Title: Phase I and Pharmacokinetic Study of Biweekly PEP02 in mCRC Refractory to 1st-line Oxaliplatin Base Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaEngine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIST-CRC-01
Record Dates: First submitted 2009-07-15; First posted 2009-07-16 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PEP02 (Experimental)
  Interventions: Drug: PEP02

INTERVENTIONS:
Drug: PEP02 — Dose escalation: 50-100 mg/m2 biweekly

SUMMARY:
The purpose of this study is to evaluate the dose-limiting toxicity (DLT), toxicity profile, maximum tolerated dose (MTD) and characterize the pharmacokinetics of biweekly PEP02 treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed metastatic colorectal cancer
* Documented disease progression after first-line chemotherapy containing oxaliplatin
* Both genders, age 18 years
* ECOG performance status 0 or 1
* Adequate organ and marrow function
* Written informed consent to participate in the study

Exclusion Criteria:

* Have received irinotecan treatment
* With active CNS metastases (indicated by clinical symptoms, cerebral edema, steroid requirement, or progressive growth)
* With clinically significant gastrointestinal disorder (e.g. bleeding, inflammation, obstruction, including partial or complete obstruction secondary to peritoneal carcinomatosis, or diarrhea > grade 1)
* With uncontrolled intercurrent illness that could limit study compliance considered to be ineligible for the study by the investigators including, but NOT limited to, any of the following:ongoing or active infection requiring antibiotic treatment, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia psychiatric illness or social situation that would preclude study compliance
* With other primary malignancies, except those remain disease-free for 3 or more years after curative treatment.
* Prior chemotherapy within 3 weeks
* Major surgery or radiotherapy within 4 weeks
* Prior participation in any investigational drug study within 3 weeks
* History of allergic reaction to liposome product
* Pregnant or breastfeeding (a urine pregnancy test must be performed on all patients who are of childbearing potential before entering the study, and the result must be negative)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2012-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the DLT and the toxicity profile | 3 years
To establish the MTD | 3 years
To characterize the pharmacokinetics of biweekly PEP02 in patients with metastatic colorectal cancer who failed to first-line oxaliplatin-based chemotherapy | 3 years

SECONDARY OUTCOMES:
To collect data for preliminary evaluation of tumor response | 3 years
To explore the association of the pharmacogenetics of PEP02 including UGT1A family - UGT1A1 and UGT1A9 with pharmacokinetic parameters and toxicity | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan